CLINICAL TRIAL: NCT05582863
Title: Effects of a 12-week Virtual Reality-based Fitness Intervention on the Functional Fitness of Adults of Different Age Ranges
Brief Title: Effects of a 12-week VR Intervention on the Functional Fitness of Adults of Different Age Ranges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: litingwang_1
Record Dates: First submitted 2022-09-23; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Functional Fitness; Virtual Reality
Keywords: Virtual reality; Exercise; Old adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group. (Experimental): The experimental group attended a VR exercise routine twice a week for 12 weeks.
  Device:1 computer virtual reality online software and 3 large projectors were used to project videos on the wall in a wrap-around state.
  Interventions: Other: Virtual reality exercise intervention
- Control group. (No Intervention): Participants in the control group received no intervention and had normal daily activites.

INTERVENTIONS:
Other: Virtual reality exercise intervention — The experimental group performed a 75-90-minute VR exercise routine twice a week for 12 weeks.
  Arms: Intervention group.

SUMMARY:
This study aimed to evaluate the effects of a 12-week VR fitness intervention on the functional fitness of adults of different age ranges.

DETAILED DESCRIPTION:
Previous studies have shown age-related decreases in physical activity and functional fitness among older adults. Virtual Reality (VR) exercise programs are currently used in leisure and entertainment to improve the physical health of older adults. However, VR exercise in assessing physical health or functional fitness in older adults of different age ranges is rare. To fill this research gap, VR exercise was to assess functional fitness improvement in young and middle-aged participants.

ELIGIBILITY:
Inclusion Criteria:

* aged more 65 and less 84 years
* with no listening/vision impairments
* who did not have any history of illness based on their response to the Physical Activity Readiness Questionnaire (PAR-Q)
* interested in the virtual reality exercise

Exclusion Criteria:

* age less than 65 or more than 84 years
* disability and unable to live independently

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-02-06 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Senior Fitness Test | Senior Functional fitness to specify a period "change" is being assessed. The time points for assessment were week 1 (pre-test), and 12 (post-test).
  The Senior Fitness Test was used to assess the functional fitness of the participants. The test has six items and evaluations of four physical functional dimensions using the following movements: Back scratch was assessed for upper body flexibility (units of measurement: cm). Chair sit-and-reach movement evaluates lower body flexibility (cm). Arm curl movement assesses upper body strength (times). Chair-stand test evaluates lower body muscle strength (times). 2-minute step exercise evaluates cardiorespiratory fitness (times). 8-foot up-and-go evaluates balance and agility, (sec).
  The back scratch, chair-and-reach, arm curl, chair stand, and 2-minute step of higher scores mean better functional fitness. The 8-foot up-and-go of higher scores means poorer functional fitness.
  The study measures the change in functional fitness of older adults from a 1-week baseline to 12 weeks (i.e., exercise intervention phase).

SECONDARY OUTCOMES:
Weight and Kilograms test | Not assessing change.The test was only a one-time measure at week 1(pre-test).
  Measure older adults of height by attaching cloth ruler tape to the wall (e.g., height in centimeters).
  The weight of the elderly is measured using commercially available electronic weighing machines. (e.g., weight in kilograms).
  The height and weight measurements of older people are aggregated to produce a reported value (e.g., weight and height will be combined to report BMI in kg/m2).

CONTACTS AND LOCATIONS:
Overall Officials: Lee Szu-Hsien, Study Director — Research Ethics Committee, National Taiwan University
Locations (1):
- NTNU, Taipei, Taiwan